CLINICAL TRIAL: NCT00305656
Title: A Phase II Study of AZD2171 in Recurrent Glioblastoma
Brief Title: AZD2171 in Treating Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00127; 05-254; N02CO12400 (Other Grant/Funding Number: US NIH Grant/Contract Award Number); CDR0000460079 (Registry Identifier: PDQ (Physician Data Query)); NCT00254943 (obsolete NCT alias)
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-07

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral AZD2171 once daily on days 1-28.
  Interventions: Drug: cediranib maleate

INTERVENTIONS:
Drug: cediranib maleate — Given orally
  Other Names: AZD2171; Recentin

SUMMARY:
This phase II trial is studying how well AZD2171 works in treating patients with recurrent glioblastoma multiforme. AZD2171 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the proportion of patients with recurrent glioblastoma multiforme (GM) who are alive and progression free 6 months after starting AZD2171 therapy.

SECONDARY OBJECTIVES:

I. Assess the biological effect of AZD2171 by using the following MRI techniques: dynamic contrast-enhanced imaging; arterial spin-labeling imaging; perfusion-weighted imaging; and diffusion- tensor imaging at serial time points.

II. Measure circulating endothelial and progenitor cells and plasma levels of tumstatin, (vascular endothelial growth factor (VEGF)-A and -D, sVEGF receptors, P1GF, platelet-derived growth factor (PDGF)-AA, PDGF-AB, PDGF-BB, Ang1, thrombospondin-1, and interleukin-8 as markers for response to antiangiogenic therapy in recurrent GM.

III. Correlate treatment outcomes with pre-AZD2171 tumor specimens with respect to microvascular density, basement membrane and pericyte coverage, and angiopoietin-1 and -2 expression to determine whether these immunohistochemical analyses can be predictive of the response to AZD2171.

IV. Measure polymorphisms of kdr/flk-1 gene and genetic analysis of HIF1-alpha, TP53, and endothelial nitric oxide synthase genes in the archival tumor specimens.

V. Determine the overall survival of patients with recurrent GM treated with AZD2171.

VI. Determine the radiographic response rate in patients with recurrent GM treated with AZD2171.

VII. Determine the safety of AZD2171 in this patient population.

OUTLINE: This is a multicenter study.

Patients receive oral AZD2171 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 12 months.

ELIGIBILITY:
Criteria:

* AST/ALT =< 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance >= 60 mL/min
* Measurable contrast-enhancing tumor >= 1 cm in longest diameter by baseline MRI or CT scan:

  * Patient must have been on no steroids OR a stable dose of steroids for >= 5 days prior to baseline MRI or CT scan
  * Patients who are on steroids must be maintained on a stable corticosteroid regimen from baseline scan until the start of study treatment
* No intratumoral or peritumoral hemorrhage by MRI
* Karnofsky performance status >= 60%
* No other concurrent malignancy within the past 5 years except curatively treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast
* Mini-mental status examination score >= 15
* Histologically confirmed glioblastoma multiforme
* Platelet count >= 100,000/mm3
* Hemoglobin >= 8 g/dL
* Bilirubin normal
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD2171
* Mean QTc =< 470 msec (with Bazett's correction) on screening electrocardiogram
* No history of familial long QT syndrome
* No greater than +1 proteinuria on 2 consecutive dipsticks taken >= 1 week apart unless first urinalysis shows no protein
* No uncontrolled intercurrent illness, including, but not limited to, any of the following:

Hypertension; Ongoing or active infection; Symptomatic congestive heart failure; Unstable angina pectoris; Cardiac arrhythmia; Psychiatric illness/social situations that would limit compliance with study requirements

* No known coagulopathy that increases the risk of bleeding
* No history of clinically significant hemorrhages
* Recovered from toxicity of prior therapy
* At least 3 months since prior radiation therapy, including cranial radiation therapy
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* At least 3 weeks since prior molecularly-targeted agents
* At least 4 weeks since prior major surgery
* No more than 2 prior chemotherapy regimens or antineoplastic drugs
* More than 30 days since prior participation in an investigational trial
* At least 2 weeks since prior enzyme-inducing antiepileptic drugs (EIAEDs)
* No concurrent EIAEDs; Concurrent non-EIAEDs allowed
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No concurrent vascular endothelial growth factor inhibitors:

Prior thalidomide or lenolidomide allowed

* No concurrent anticoagulants (e.g., warfarin) or antiplatelet agents including aspirin
* No other concurrent anticancer agents or therapies
* No concurrent grapefruit juice
* WBC >= 3,000/mm3
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Absolute neutrophil count >= 1,500/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-01; Primary Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients alive and progression-free at 6 months | 6 months

SECONDARY OUTCOMES:
Radiographic response proportion | Up to 12 months
  Will be described with 95% confidence limits.
Overall survival | Up to 12 months
  Will be described with 95% confidence limits.
Toxicity proportion | Up to 12 months
  Will be described with 95% confidence limits.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Batchelor, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Batchelor TT, Duda DG, di Tomaso E, Ancukiewicz M, Plotkin SR, Gerstner E, Eichler AF, Drappatz J, Hochberg FH, Benner T, Louis DN, Cohen KS, Chea H, Exarhopoulos A, Loeffler JS, Moses MA, Ivy P, Sorensen AG, Wen PY, Jain RK. Phase II study of cediranib, an oral pan-vascular endothelial growth factor receptor tyrosine kinase inhibitor, in patients with recurrent glioblastoma. J Clin Oncol. 2010 Jun 10;28(17):2817-23. doi: 10.1200/JCO.2009.26.3988. Epub 2010 May 10. PMID 20458050
- [Derived] Emblem KE, Farrar CT, Gerstner ER, Batchelor TT, Borra RJ, Rosen BR, Sorensen AG, Jain RK. Vessel caliber--a potential MRI biomarker of tumour response in clinical trials. Nat Rev Clin Oncol. 2014 Oct;11(10):566-84. doi: 10.1038/nrclinonc.2014.126. Epub 2014 Aug 12. PMID 25113840